CLINICAL TRIAL: NCT06653608
Title: Clinical Efficacy of Novel Jasminum-based Nano-reinforced Calcium Hydroxide Medicament on Postoperative Pain: a Triple-blind Study
Brief Title: Clinical Efficacy of Novel Jasminum-based Calcium Hydroxide Medicament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, NEHAL AMIR, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOD/ERB/2024/58
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Necrotic Pulp; Acute Apical Periodontitis of Pulpal Origin
Keywords: Endodontic; Necrotic pulp; Apical Periodontitis
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this triple-blind trial, participants, care provider and outcome assessor were unaware of the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Nano-reinforced Calcium hydroxide) (Experimental): Nano-reinforced Calcium hydroxide Medicament
  Interventions: Drug: Nano-reinforced calcium hydroxide medicament
- Group B (Conventional Calcium hydroxide) (Experimental): Calcium hydroxide without nanoparticles
  Interventions: Drug: Calcium hydroxide without nanoparicles

INTERVENTIONS:
Drug: Nano-reinforced calcium hydroxide medicament — Group A (Calcium hydroxide intracanal medicament reinforced with jasminum derived- titania nanoparticles)
  Other Names: Group A
  Arms: Group A (Nano-reinforced Calcium hydroxide)
Drug: Calcium hydroxide without nanoparicles — Group B ( Calcium hydroxide medicament without nanoparticles)
  Other Names: Group B
  Arms: Group B (Conventional Calcium hydroxide)

SUMMARY:
A triple-blind, parallel group, randomized trial with an allocation ratio of 1:1. Participants randomly allocated into two groups A and B. In group A, nano-reinforced calcium hydroxide medicament was utilized while in group B, calcium hydroxide medicament without nanoparticles was used. Post-operative pain was assessed after 4 hours, 24 hours, 48 hours, 72 hours, 96 hours.

DETAILED DESCRIPTION:
This triple-blind parallel group, randomized clinical trial was conducted at the department of Operative Dentistry and Endodontics, School of Dentistry from April 24, 2024 to September 25, 2024. Participants were randomly distributed into two groups by Lottery method. A consecutive non-probability sampling technique was used. Before initiating treatment, participants were briefed about the intervention and their preoperative pain score was recorded. In both groups, endodontic treatment was initiated under rubber dam isolation. Access opening done and canals explored. Working length taken by radiographic method and reconfirmed by an electronic apex locator. Afterwards, canals were prepared till Master Apical File size F2 (4% Taper). In group A, Nano-reinforced calcium hydroxide medicament was placed while in group B, calcium hydroxide without nanoparticles was utilized. Participants were instructed to rate their postoperative pain record after 4hrs, 24hrs, 48hrs, 72hrs and 96hrs.

ELIGIBILITY:
Inclusion Criteria:

* Participants with good general health status
* Necrotic pulp with Symptomatic Apical Periodontitis
* Single rooted teeth

Exclusion Criteria:

* Non-restorable teeth
* Teeth associated with acute or chronic apical abscess
* Teeth with chronic periodontitis
* Teeth with anatomical complexities or complications like open apex, calcified canal, severe root dilaceration, root resorptive defects
* Participants who received antibiotic treatment during the last 3 months
* Pregnant females
* Participants on pre-treatment analgesics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | One week
  Pain scores assessed by Visual Analogue Scale (VAS) score after 4hr, 24hrs, 48hrs, 72hrs, 96hrs. The minimum score is O (None) and the maximum score is 10 (Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Amir, BDS, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AM, Gangoo IKA, Ali NA, Khan M, Javed MQ, AlAttas MH, Abulhamael AM, Bahammam HA, Alsofi L, Yahya RSA. The Effect of Calcium Hydroxide, Triple Antibiotic Paste and Chlorhexidine on Pain in Teeth with Symptomatic Apical Periodontitis: A Randomised Controlled Trial. Int J Environ Res Public Health. 2023 Feb 10;20(4):3091. doi: 10.3390/ijerph20043091. PMID 36833788
- [Background] Ghanbarzadegan A, Ajami M, Aminsobhani M. The Effect of Different Combinations of Calcium Hydroxide as Intra-Canal Medicament on Endodontic Pain: A Randomized Clinical Trial Study. Iran Endod J. 2019 Winter;14(1):1-6. doi: 10.22037/iej.v14i1.22815. PMID 36879602
- [Derived] Amir N, Mansoor E, Eeman N, Ahmed MN, Mansoor E, Mansoor E, Hussain K, Afreixo V, Mansoor A, Brochado Martins JF, Palma PJ. Jasminum-based Nano-reinforced Calcium Hydroxide Reduces Postoperative Pain in Symptomatic Apical Periodontitis: A Randomized Controlled Trial. J Endod. 2025 Aug;51(8):996-1005. doi: 10.1016/j.joen.2025.05.016. Epub 2025 Jun 2. PMID 40466913